CLINICAL TRIAL: NCT03592095
Title: Blinding of Dry Needling Technique Based on Previous Experiences: A Double-blinded Clinical Trial
Brief Title: Blinding and Previous Experiences of Dry Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Gracia Gallego Sendarrubias, Proffesor, European University of Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hulp:5006
Record Dates: First submitted 2018-06-02; First posted 2018-07-19 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Neck Pain
Keywords: Dry needling; Placebo; Myofascial pain syndrome; Blinding
MeSH Terms: conditions — Neck Pain; Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DN group (Experimental): The intervention group will receive real dry needling (DN) (fast in and fast out needling technique) in an active MTrP within upper trapezius muscle.
  Interventions: Device: Dry needling
- Placebo needle (Placebo Comparator): The placebo group will receive sham needling in an active MTrP within the upper trapezius muscle. A sham needle will be used as placebo. This needle has a blunt tip and retractable handle that created the illusion of a needle penetrating the skin.
  Interventions: Device: Placebo needle

INTERVENTIONS:
Device: Dry needling — Real dry needling will be conducted according to Hong description, fast-in and fast-out interventions. The intervention will be applied until a total of four local twitch responses will be elicited
  Arms: DN group
Device: Placebo needle — Sham dry needling with be conducted with a sham needle (Steitberger's Park sham device (PSD). This needle has a blunt tip and retractable handle that created the illusion of a needle penetrating the skin. When this needle touches the skin, a pricking sensation will be created. However, when pressure will be increased, the shaft of the needle disappears into the handle creating a sensation on the patient.
  Arms: Placebo needle

SUMMARY:
Dry needling (DN) is a treatment technique widely used in patients with various musculoskeletal health problems due to myofascial trigger points (MTrP). DN has shown to have positive effect on pain and function in patients with mechanical neck pain. These positive results are thought to be the consequence of specific neurophysiological and mechanical processes. Research has shown that DN induces 1) end plate inhibition, 2) reduction of inflammatory substances, 3) increase of blood flow and oxygen and 4) a reduction of nociceptive afferent activity. However, the exact working mechanisms underlying DN effects is still a topic of debate. This trial addresses one of the major methodological issues in needle testing,the effects of proper blinding. DN is a specific technique that is not easily be replaced by another comparable intervention. A sham needle with a blunt tip was created that simulates penetration into the skin without actually doing so. Research about a valid method for the control in needling studies is for this reason of particular relevance. A proper blinding technique is of importance to further the field of DN.

DETAILED DESCRIPTION:
The objectives of this study are to analysize short-term effects on pain intensity and pressure pain sensitivity according to previous experience (blinding) in subjects with mechanical neck pain receiving real or sham-DN and to determine the success in masking DN versus sham DN in patients with mechanical neck pain based on prior experience with this technique.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific mechanical neck pain of at least 3 months of duration
* Between 18-60 years old
* At least one active trigger point in the upper trapezius muscle which referred pain reproduces the neck pain symptoms

Exclusion Criteria:

* whiplash injury;
* previous cervical or thoracic surgery;
* cervical radiculopathy or myelopathy;
* diagnosis of fibromyalgia syndrome;
* having undergone physical therapy in the previous 6 months;
* fear to needles

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Changes in Neck Pain Intensity between baseline and follow-up periods | Baseline, inmediately after and 1 week after intervention
  The intensity of neck pain at rest and during active movement of the cervical spine in rotation will be assessed with a visual analogue scale (VAS).
Identification (blinding) of the needling intervention | Inmediately after intervention
  Participants will be asked directly after the intervention whether they thought they had received a real intervention or a sham. Answering categories were: 'yes' (real DN) or 'no' (sham DN).

SECONDARY OUTCOMES:
Changes in Pressure pain sensitivity between baseline and follow-up periods | Baseline, inmediately after and 1 week after intervention
  Pressure pain thresholds (PPT) will be assessed at the upper trapezius muscle, spinous process of C7 and distant pain-free area of the lower extremity (heel)
Changes in patients self-perceived improvement between baseline and follow-up periods | Baseline and 1 week after intervention
  Patients self-perceived improvement will be assessed using a Global Rating of Change (GROC) consisting of a 15-point scale ranging from -7 (a very great deal worse) to +7 (a very great deal better).
  Descriptors of worsening or improving are assigned with values ranging from -1 to -7 and +1 to +7, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Gracia Gallego-Sendarrubias, Madrid, Rest of the World, Spain